CLINICAL TRIAL: NCT04414202
Title: Observational Study of Intra-operative Partial Irradiation of Invasive Ductal Breast Carcinomas With a Good Prognosis
Acronym: INTRA-OBS
Status: Active, not recruiting | Type: Observational
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/OBS-01
Record Dates: First submitted 2020-05-19; First posted 2020-06-04 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Invasive Breast Cancer; Breast-conserving Surgery
Keywords: breast cancer; good prognosis; surgery; intra-operative partial irradiation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 GROUP: Patient with an Invasive breast cancer with a good prognosis that is accessible to breast-conserving surgery.
  The treatment combines extended tumorectomy with axillary dissection (sentinel lymph node) in addition to 20 Gy of per-operative partial irradiation at the tumor Follow up after this treatment will scheduled 10 years
  Interventions: Procedure: tumorectomy with axillary dissection (sentinel lymph node); Radiation: per-operative partial irradiation

INTERVENTIONS:
Procedure: tumorectomy with axillary dissection (sentinel lymph node) — All patients will have local excision of the primary tumor following appropriate clinical work-up. Surgery will be done according to usual local practice with a complete excision of the tumor. The aim of the local excision should be to achieve a minimum free margin of 2 mm whilst maintaining a good cosmetic outcome.
Radiation: per-operative partial irradiation — 20 Gy of per-operative partial irradiation at the tumor site during the surgery

SUMMARY:
Due to screening, T1N0 early-stage breast cancer now accounts for more than 50% of the tumors diagnosed in France. The prognosis of these tumors is good, even excellent in women ≥ 65 years of age, with specific survival of 98% at 5 years.

The treatment of these tumors combines breast-conserving surgery and external whole breast irradiation for 6.5 weeks.

A true de-escalation of treatment is taking place with these tumors, both surgically and medically. Surgery therefore now prefers breast-conserving methods in combination with exeresis of the sentinel lymph node only. In the same way, in many international studies, radiotherapy has been evaluating the possibility of reducing both:

* the irradiation volume at the excision site (partial irradiation)
* the duration of this irradiation (accelerated radiotherapy)

Between 2004 and 2007, the CRLC [Regional Anti-Cancer Center] evaluated the feasibility and the oncological results of intra-operative partial irradiation via a phase II study in women 65 years of age and older with T1N0M0 hormone-sensitive tumors with a good prognosis.

From 2010 to 2013, the ICM carried out an observational study of these tumors with an excellent prognosis.

In July 2009, the American Society for Radiation Oncology (ASTRO) published a consensus statement with specific recommendations and indications for accelerated partial breast irradiation (APBI).

This APBI technique has been developing in France over the past 5 years within the framework of clinical studies and in compliance with the 2012 recommendations of the French National Cancer Institute. This APBI can be given by 3D external radiotherapy or, as in this study, by intra-operative radiotherapy (IORT) in order to obtain optimal precision and spare as much of the surrounding healthy tissue as possible.

The Investigator therefore propose a cohort study to prospectively analyze the results of this technique applied to the indications strictly defined by the ASTRO.

DETAILED DESCRIPTION:
after registration, particpants have as treatment "combination extended tumorectomy with axillary dissection (sentinel lymph node) in addition to 20 Gy of per-operative partial irradiation at the tumor site.

follow up after this treatment during 5 years

ELIGIBILITY:
Inclusion Criteria:

* Women 60 years of age or older,
* Histologically proven invasive ductal breast cancer or of a histologically favorable sub-type (mucinous, tubular or colloid),

  -. Unifocal tumor,
* T1 (diameter ≤ 20 mm),
* N0 (pN0 or pNi+),
* M0,
* Gland exeresis margins ≥ 2 mm,
* Estrogen receptor positive,
* Information and non-opposition of the patient.

Exclusion Criteria:

-. Inflammatory breast cancer,

* Associated peri-tumoral lymphatic emboli
* Associated extensive intra-ductal component
* Invasive lobular carcinoma
* Pure ductal carcinoma in situ,
* Sarcoma or lymphoma-type non-epithelial tumor
* Synchronous bilateral breast cancer,
* Any prior neo-adjuvant treatment: radiotherapy, chemotherapy, hormone therapy

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Invasive breast cancer with a good prognosis that is accessible to breast-conserving surgery
Sampling Method: Probability Sample
Enrollment: 519 (Actual)
Dates: Start 2009-12-15 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2030-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: LEMANSKI Claire, DR, Study Chair — ICM Val d'Aurelle DRCI
Locations (1):
- Icm Val D'Aurelle, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grosclaude P, Colonna M, Hedelin G, Tretarre B, Arveux P, Lesec'h JM, Raverdy N, Sauvage-Machelard M. Survival of women with breast cancer in france: variation with age, stage and treatment. Breast Cancer Res Treat. 2001 Nov;70(2):137-43. doi: 10.1023/a:1012974728007. PMID 11768604
- [Background] van Dongen JA, Voogd AC, Fentiman IS, Legrand C, Sylvester RJ, Tong D, van der Schueren E, Helle PA, van Zijl K, Bartelink H. Long-term results of a randomized trial comparing breast-conserving therapy with mastectomy: European Organization for Research and Treatment of Cancer 10801 trial. J Natl Cancer Inst. 2000 Jul 19;92(14):1143-50. doi: 10.1093/jnci/92.14.1143. PMID 10904087
- [Background] Veronesi U, Cascinelli N, Mariani L, Greco M, Saccozzi R, Luini A, Aguilar M, Marubini E. Twenty-year follow-up of a randomized study comparing breast-conserving surgery with radical mastectomy for early breast cancer. N Engl J Med. 2002 Oct 17;347(16):1227-32. doi: 10.1056/NEJMoa020989. PMID 12393819
- [Background] Clarke M, Collins R, Darby S, Davies C, Elphinstone P, Evans V, Godwin J, Gray R, Hicks C, James S, MacKinnon E, McGale P, McHugh T, Peto R, Taylor C, Wang Y; Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of radiotherapy and of differences in the extent of surgery for early breast cancer on local recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 Dec 17;366(9503):2087-106. doi: 10.1016/S0140-6736(05)67887-7. PMID 16360786
- [Background] Bartelink H, Horiot JC, Poortmans PM, Struikmans H, Van den Bogaert W, Fourquet A, Jager JJ, Hoogenraad WJ, Oei SB, Warlam-Rodenhuis CC, Pierart M, Collette L. Impact of a higher radiation dose on local control and survival in breast-conserving therapy of early breast cancer: 10-year results of the randomized boost versus no boost EORTC 22881-10882 trial. J Clin Oncol. 2007 Aug 1;25(22):3259-65. doi: 10.1200/JCO.2007.11.4991. Epub 2007 Jun 18. PMID 17577015
- [Background] Dubois JB, Hay M, Gely S, Saint-Aubert B, Rouanet P, Pujol H. IORT in breast carcinomas. Front Radiat Ther Oncol. 1997;31:131-7. doi: 10.1159/000061160. No abstract available. PMID 9263806
- [Background] Lemanski C, Azria D, Thezenas S, Gutowski M, Saint-Aubert B, Rouanet P, Fenoglietto P, Ailleres N, Dubois JB. Intraoperative radiotherapy given as a boost for early breast cancer: long-term clinical and cosmetic results. Int J Radiat Oncol Biol Phys. 2006 Apr 1;64(5):1410-5. doi: 10.1016/j.ijrobp.2005.10.025. Epub 2006 Jan 25. PMID 16442241
- [Background] Lemanski C, Azria D, Gourgon-Bourgade S, Gutowski M, Rouanet P, Saint-Aubert B, Ailleres N, Fenoglietto P, Dubois JB. Intraoperative radiotherapy in early-stage breast cancer: results of the montpellier phase II trial. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3):698-703. doi: 10.1016/j.ijrobp.2009.02.039. Epub 2009 May 23. PMID 19467579
- [Background] Smith BD, Arthur DW, Buchholz TA, Haffty BG, Hahn CA, Hardenbergh PH, Julian TB, Marks LB, Todor DA, Vicini FA, Whelan TJ, White J, Wo JY, Harris JR. Accelerated partial breast irradiation consensus statement from the American Society for Radiation Oncology (ASTRO). J Am Coll Surg. 2009 Aug;209(2):269-77. doi: 10.1016/j.jamcollsurg.2009.02.066. Epub 2009 Apr 24. No abstract available. PMID 19632605
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Background] Vlastos G, Mirza NQ, Meric F, Hunt KK, Kuerer HM, Ames FC, Ross MI, Buchholz TA, Hortobagyi GN, Singletary SE. Breast conservation therapy as a treatment option for the elderly. The M. D. Anderson experience. Cancer. 2001 Sep 1;92(5):1092-100. doi: 10.1002/1097-0142(20010901)92:53.0.co;2-p. PMID 11571720
- [Background] Vinh-Hung V, Verschraegen C. Breast-conserving surgery with or without radiotherapy: pooled-analysis for risks of ipsilateral breast tumor recurrence and mortality. J Natl Cancer Inst. 2004 Jan 21;96(2):115-21. doi: 10.1093/jnci/djh013. PMID 14734701
- See also: Institut de Veille Sanitaire- Institut National du Cancer — https://www.e-cancer.fr/

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 GROUP: Patient with an Invasive breast cancer with a good prognosis that is accessible to breast-conserving surgery.
  The treatment combines extended tumorectomy with axillary dissection (sentinel lymph node) in addition to 20 Gy of per-operative partial irradiation at the tumor Follow up after this treatment will scheduled 10 years
  tumorectomy with axillary dissection (sentinel lymph node): All patients will have local excision of the primary tumor following appropriate clinical work-up. Surgery will be done according to usual local practice with a complete excision of the tumor. The aim of the local excision should be to achieve a minimum free margin of 2 mm whilst maintaining a good cosmetic outcome.
  per-operative partial irradiation: 20 Gy of per-operative partial irradiation at the tumor site during the surgery
Period: Overall Study
Arm/Group | 1 GROUP
Started | 519
Completed | 496
Not Completed | 23

BASELINE CHARACTERISTICS:
Arm/Group | 1 GROUP
Number analyzed (Participants) | 519
Age, Continuous [Mean (Full Range); unit: years] | 69.54 [59 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 519
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patient With a Local Intra-mammary Relapse
Description: The local relapse rate, defined as the number of intramammary relapses in the treated breast (regardless of quadrant and including skin), appreciated at 5 years and 10 years. It will be assessed according to the recommendations applied to the Centre
Time Frame: post surgery : 3 weeks, every 6 months during 5 years and annually during 5 years (10 years in total)
Measure: Count of Participants; unit: Participants
Arm/Group | 1 GROUP
Number analyzed (Participants) | 519
Participants
  no relapse | 498
  local relapse | 15
  local and metastatic relapse | 1
  not specified | 5

2. Secondary Outcome: Cosmetic Results
Description: Evaluation of the cosmetic result of questionnaire (0 "no satisfy with the cosmetic result"" from 10 "very satisfy with the cosmetic result")
Time Frame: post surgery : 3 weeks, 6 months and 12 months
Population: the number of patient wich respond to the cosmetic questionnaire differs from the Overall Number of Participants Analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | 1 GROUP
Number analyzed (Participants) | 519
Participants
  at 3 weeks after the treatment: very good cosmetic result | 208
  at 3 weeks after the treatment: good cosmetic result | 124
  at 3 weeks after the treatment: bad cosmetic result | 12
  at 3 weeks after the treatment: very bad cosmetic result | 0
  at 3 weeks after the treatment: no data | 175
  at 6 months after the treatment: very good cosmetic result | 198
  at 6 months after the treatment: good cosmetic result | 147
  at 6 months after the treatment: bad cosmetic result | 14
  at 6 months after the treatment: very bad cosmetic result | 1
  at 6 months after the treatment: no data | 159
  at 12 months after the treatment: very good cosmetic result | 256
  at 12 months after the treatment: good cosmetic result | 99
  at 12 months after the treatment: bad cosmetic result | 9
  at 12 months after the treatment: very bad cosmetic result | 1
  at 12 months after the treatment: no data | 154

3. Secondary Outcome: Patients' Satisfaction Towards the Treatment
Description: Satisfaction will be measured using the Likert scale (0 no satisfy to 10: strongly satisfy)
Time Frame: post surgery : 3 weeks, 6 months and 12 months
Population: patient no completed the Likert scale
Measure: Count of Participants; unit: Participants
Arm/Group | 1 GROUP
Number analyzed (Participants) | 519
Participants
  At 3 weeks after the treatment: number analyzed (Participants) | 516
  At 3 weeks after the treatment: Very good satisfaction | 135
  At 3 weeks after the treatment: good satisfaction | 200
  At 3 weeks after the treatment: bad satisfaction | 30
  At 3 weeks after the treatment: very bad satisfaction | 1
  At 3 weeks after the treatment: missing | 150
  At 6 months after the treatment: number analyzed (Participants) | 481
  At 6 months after the treatment: Very good satisfaction | 165
  At 6 months after the treatment: good satisfaction | 198
  At 6 months after the treatment: bad satisfaction | 20
  At 6 months after the treatment: very bad satisfaction | 1
  At 6 months after the treatment: missing | 97
  At 12 months after the treatment: number analyzed (Participants) | 461
  At 12 months after the treatment: Very good satisfaction | 173
  At 12 months after the treatment: good satisfaction | 188
  At 12 months after the treatment: bad satisfaction | 26
  At 12 months after the treatment: very bad satisfaction | 3
  At 12 months after the treatment: missing | 71

4. Secondary Outcome: Impact of the Accelerated Treatment on the Maintenance of Autonomy in Elderly Patients
Description: Assessment of the impact of this accelerated treatment on maintaining the autonomy of the subject by the use of geriatric scale (ADL (Activities of Daily Living), IADL (instrumental Activities of Daily Living)). (scale from 0 "no autonomy" to 10 "good autonomy")
Time Frame: post surgery : 3 weeks, 6 months and 12 months
Population: patient no completed scale with the time
Measure: Count of Participants; unit: Participants
Arm/Group | 1 GROUP
Number analyzed (Participants) | 519
Participants
  At 3 weeks post treatment: number analyzed (Participants) | 516
  At 3 weeks post treatment: 0 "no autonomy" | 1
  At 3 weeks post treatment: 3 | 1
  At 3 weeks post treatment: 4 | 0
  At 3 weeks post treatment: 5 | 7
  At 3 weeks post treatment: 6 | 5
  At 3 weeks post treatment: 7 | 7
  At 3 weeks post treatment: 8 | 36
  At 3 weeks post treatment: 9 | 67
  At 3 weeks post treatment: 10 "good autonomy" | 246
  At 3 weeks post treatment: Missing | 146
  At 6 months post treatment: number analyzed (Participants) | 481
  At 6 months post treatment: 0 "no autonomy" | 0
  At 6 months post treatment: 3 | 0
  At 6 months post treatment: 4 | 1
  At 6 months post treatment: 5 | 9
  At 6 months post treatment: 6 | 2
  At 6 months post treatment: 7 | 10
  At 6 months post treatment: 8 | 41
  At 6 months post treatment: 9 | 65
  At 6 months post treatment: 10 "good autonomy" | 256
  At 6 months post treatment: Missing | 97
  At 12 months post treatment: number analyzed (Participants) | 461
  At 12 months post treatment: 0 "no autonomy" | 0
  At 12 months post treatment: 3 | 1
  At 12 months post treatment: 4 | 1
  At 12 months post treatment: 5 | 3
  At 12 months post treatment: 6 | 3
  At 12 months post treatment: 7 | 15
  At 12 months post treatment: 8 | 42
  At 12 months post treatment: 9 | 72
  At 12 months post treatment: 10 "good autonomy" | 250
  At 12 months post treatment: Missing | 74

5. Secondary Outcome: Overall Survival
Description: rate of death
Time Frame: from baseline to 10 years after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 1 GROUP
Number analyzed (Participants) | 519
Participants
  Alive | 441
  deceased | 39
  lost of follow up | 39

ADVERSE EVENTS:
Time Frame: collection from the baseline to 120 months after treatment by radiotherapy
Description: adverse event collected with CTCAE. no serious adverse event appeared
Arm/Group | 1 GROUP
All-Cause Mortality (participants affected / at risk) | 39/519
Serious Adverse Events (participants affected / at risk) | 0/519
Other Adverse Events (participants affected / at risk) | 519/519
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 GROUP (N=519)
atrophy (General disorders) | 14 (14) — atrophy grade 1 or 2
cutaneous eruption (General disorders) | 3 (3) — cutaneous eruption grade 1
fibrosis (Musculoskeletal and connective tissue disorders) | 383 (383) — fibrosis grade 1, 2
hyperpigmentation (Musculoskeletal and connective tissue disorders) | 97 (97) — hyperpigmentation grade 1 and 2
erythema redness (Musculoskeletal and connective tissue disorders) | 38 (38) — erythema redness grade 1 and 2
telangiectasia (Musculoskeletal and connective tissue disorders) | 13 (13) — telangiectasia grade 1
ulceration (Musculoskeletal and connective tissue disorders) | 4 (4) — ulceration grade 1 and 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2009-12-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT04414202/Prot_000.pdf